CLINICAL TRIAL: NCT04679922
Title: Fascia Lata Allograft Versus Subepithelial Connective Tissue Grafts in the Peri-Implant
Brief Title: Fascia Lata Allograft Versus Subepithelial Connective Tissue Grafts in the Peri-Implant Mucosal Thickness Enhancement.
Acronym: Fascia Lata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Hamdy Helal (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Hamdy Helal, Assistant Professor Malak Yousef Mohamed Shoukheba, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMPDR-07-19-5
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Implant Tissue Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri Implant mucosal thickness connective tissue graft (Active Comparator)
  Interventions: Procedure: Soft Tissue Enhancement around dental implant
- Peri Implant mucosal thickness fascia lata graft (Experimental)
  Interventions: Procedure: Soft Tissue Enhancement around dental implant

INTERVENTIONS:
Procedure: Soft Tissue Enhancement around dental implant — Sixteen sites that are indicated for peri-implant mucosal augmentation at the time of implant placement will be selected. Sixteen sites that were met the subsequent inclusion criteria were eligible to contribute in our study were classified randomly by the sealed envelope technique into two treatment groups, 8 sites in each group. Group I (Control Group): Autogenous SCTGs harvested from the palate +dental implants *. Group II (Experimental Group): FLA **+dental implants. The allocation was withheld from the surgeon (M.H.) until just before the surgical appointment. The clinical examiner (M.S.) was masked to the treatment group for the extent of the study.Three months after implantation, the sites were located, and the thickness of the mucosa will be evaluated using the customized stent. The operculectomy will be performed following the method of Flatebo et al.,22 collecting biopsy specimens of almost constant quality and evaluating clinical thickness without mucosal distortions

SUMMARY:
The aim of this, randomized clinical trial is to determine the clinical efficacy of fascia lata allograft in terms of peri-implant mucosal augmentation, as compared to autologous sub epithelial connective tissue graft, clinically and histologically in human adults .

DETAILED DESCRIPTION:
The aim of this, randomized clinical trial is to determine the clinical efficacy of fascia lata allograft in terms of peri-implant mucosal augmentation, as compared to autologous sub epithelial connective tissue graft, clinically and histologically in human adults .

The hypothesis of the study is that a similar gain in peri implant mucosal thicknesses will be obtained in sites treated by either a sub epithelial connective tissue graft or a newly developed fascia lata allograft in clinically and histologically in human.

The objective of this study will be to evaluate the efficacy of the peri-implant mucosal thickness enhancement following either subepithelial connective tissue grafts or human Fascia Lata Allograft placed simultaneously with dental implant placement.

Sixteen sites that are indicated for peri-implant mucosal augmentation at the time of implant placement will be selected. Participants will be randomized to the control (simultaneous SCTGs) or test (simultaneous FLA) group.

ELIGIBILITY:
Inclusion Criteria:

Ability to maintain good oral hygiene as evidenced in recall visits. Aged 30 to 55 years. Stable periodontal condition and missing one single tooth (maxillary anterior teeth and premolars) with adjacent teeth present and thin mucosal phenotype (< 2mm bucco- lingual thickness).

Exclusion Criteria:

Uncontrolled diabetes mellitus. Females who were pregnant, or attempting to become pregnant, and nursing mothers.

Acute infection in the area intended for implant placement.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Peri-Implant Mucosal Thickness | Measure changes in mucosal thickness around dental implant at base line and after 6 months.
  The primary outcome of interest will be to measure changes (in mm) in horizontal PMT on the buccal aspect of the edentulous alveolar ridge from baseline (implant placement and grafting) to (4, 8, 12, and 24 weeks) of post-surgical healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No